CLINICAL TRIAL: NCT03685370
Title: PERiX: Comparison of Efficacy Between Placement of Epidural Catheters X-ray Guided and LOS Technique: Outcome Influence on Patient Underwent Pancreatic Surgery
Brief Title: PERiX: Comparison of Efficacy Between Placement of Epidural Catheters X-ray Guided and LOS Technique
Acronym: PERiX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Alvise Martini, MD, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PERiX
Record Dates: First submitted 2018-06-27; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Postoperative Pain; Postoperative Complications; Pancreatic Cancer; Haemodynamic Instability
Keywords: Epidural catheter; postoperative pain; LOS
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOS group (Active Comparator): Patients randomized to recieve epidural catheter placement with LOS technique, without any Rx control
  Interventions: Procedure: LOS
- X-ray group (Experimental): Patients randomized for X-ray placement of epidural catheter
  Interventions: Procedure: X-ray placement

INTERVENTIONS:
Procedure: LOS — placement of epidural catheters with LOS technique
  Arms: LOS group
Procedure: X-ray placement — placement of epidural catheters with x-ray guide
  Arms: X-ray group

SUMMARY:
The use of epidural catheters for postoperative analgesia in pancreatic surgery is recommended by the guidelines of the ERAS society. Some studies claim it may expose to hemodynamic alterations that may compromise outcome and increase postoperative complications, attributable to a malfunction of the catheter itself, often linked to a bad positioning, since this is usually positioned with LOS technique. Our hypothesis is that a positioning made using the radiographic guide the day before the intervention can significantly reduce the number of catheter's dysfunctions.

DETAILED DESCRIPTION:
About 30% of epidural catheters are reported to have hypo or hyper functioning behaviour. This has and impact on postoperative pain control and can affect also surgical and global outcome since it is known that a malfunctional catheter carries an increased complication's rate.

Our hypothesis is that rx-guided positioning can reduce the incidence of catheter malfunction afrom 30 to 15 %.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for open pancreatic surgery
* ASA < = 3

Exclusion Criteria:

* scoliosis
* coagulation abnormalities
* antiplatelet drugs (except ASA)
* history of back surgery
* anticipated need of ICU stay

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of catheters malfunctions in LOS and X-ray group | every day until 7th postoperative day
  malfunctional catheters are defined as following:
  * symptomatic hypotension due to epidural infusion
  * NRS > 6 in the first postoperative day and NRS > 4 in subsequent postoperative day
  * overt malpositioning:
  * rx evidence of catheter's tip under T10 during routine rx or TC
  * NRS > 6 (due to pain at T7-10 dermatomers) with 5 cc/h catheter infusion and response to lidocaine 1% 6ml bolus (low tip)
  * NRS > 6 (due to pain at T7-10 dermatomers) with 5 cc/h catheter infusion and NO response to lidocaine 1% 6ml bolus ( not in epidural space or very low tip)
  * evidence of catheter accidental removal
  Numerical Rating Scale (NRS) is used to assess pain. Patients self-report actual pain on 0 to 10 scale where 0 is no pain and 10 is the worst immaginable pain.

SECONDARY OUTCOMES:
Evaluate daily pain differences between groups: NRS (Numeric rating scale) | every day until 7th postoperative day
  Parameter used
  -higher postoperative daily numeric rating scale (NRS) until catheter removal
  Numerical Rating Scale (NRS) is used to assess pain. Patients self-report actual pain on 0 to 10 scale where 0 is no pain and 10 is the worst immaginable pain.
Monitoring postoperative surgical complications between groups | at 30th postoperative day
  Complications are considered as:
  * bleedings
  * infections
  * pancreatic fistulas (degree)
  * biliary fistulas
  * abdominal collections
  * ICU admission
  * needs of new surgery (for any reasons)
  * pneumonia
  * delayed gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Alvise Martini, MD, Principal Investigator — AOUI Verona
Locations (1):
- Azienda ospedaliero-universitaria integrata Verona, Verona, Veneto, Italy